CLINICAL TRIAL: NCT01900912
Title: Evaluating the Impact of Community Led Total Sanitation in Mali. A Randomized Controlled Trial
Brief Title: Evaluating the Impact of Community Led Total Sanitation Programs in Mali
Acronym: CLTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de La Plata (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); UNICEF (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Maria Laura Alzua, Principal Investigator - Prof, Universidad Nacional de La Plata
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GDGOPP1024012
Record Dates: First submitted 2013-03-12; First posted 2013-07-17 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Diarrhea; Respiratory Infection
Keywords: sanitation; diarrhea prevalence; health; social networks; cooperation
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLTS communities (Experimental): Assigned to a community led total sanitation (CLTS) intervention, carried out by the government with support from Unicef (n=60 communities). The CLTS intervention includes a triggering session facilitated by the government to encourage community members to build their own latrines and stop open defecation. Regular monitoring is conducted by government program staff until the community is declared open defecation free.
  Interventions: Other: CLTS
- Rural communities (No Intervention): No intervention will be delivered (n=61 communities)

INTERVENTIONS:
Other: CLTS — The goal of CLTS is to obtain Open Defecation Free (ODF) villages. CLTS aims to trigger the community's desire for change, propel them into action and encourage innovation, mutual support and appropriate local solutions, in order to foster greater ownership and sustainability. The phases are: pre-triggering (a group of trained-CLTS people visit the community and request a date to discuss sanitation-related issues for the following days), triggering (people are made to express their views on sanitation issues and their needs), monitoring (involves visits of the community twice a week for a period of 1-3 months) and certification (an external committee evaluates the village for certification as an ODF community).
  Other Names: Community Led Total Sanitation
  Arms: CLTS communities

SUMMARY:
Behavioral change is a key ingredient for successful adoption of better sanitation practices in rural Africa. Sanitation programs have, for some time now, incorporated the need to raise awareness and emphasize the benefits of toilet usage. These endeavors, often combined with subsidies linked to toilet construction by households, seek to create a demand for sanitation goods. Yet, progress in securing the desired outcomes from sanitation programs has been slow. Moreover, benefits of sanitation largely take the form of externalities, which individuals do not take into account when making their own decisions about investments. This makes sanitation promotion at the household level particularly challenging.

A new approach to sanitation entails a shift away from the provision of subsidies for toilets to individual households and a promotion of behavioral change at individual-level towards emphasizing collective decision-making in order to produce 'open defecation-free' villages. The objective of the intervention is to reduce the incidence of diseases related to poor sanitation and manage public risks posed by the failure to safely confine the excreta of some community members. The way to achieve this objective is by empowering communities motivated to take collective action. Local governments and other agencies perform a facilitating role. There is a growing recognition that this approach, referred to as Community-Led Total Sanitation (CLTS), may help with the reduction of open defecation practices. However, no rigorous impact evaluation of CLTS has been conducted so far. This randomized controlled trial will study the effect of CLTS in rural Mali. As a result, sound evidence will become available to see to what extent CLTS improves health outcomes and what is driving collective action in order to increase sanitation coverage.

The direct recipients of the intervention are members of rural communities in Mali who aspire to live in a cleaner environment. The donor community, international organizations, and governments in developing countries will benefit from having simple and clear evidence on the effectiveness of an innovative program for improving sanitation in rural areas. They will learn whether the program has worked or failed to achieve its objective of eradicating open defecation, and about key factors explaining success and failure.

DETAILED DESCRIPTION:
The evaluation study described involves 121 communities in the Region of Koulikoro in rural Mali. The intervention works in the following manner: communities are facilitated (by means of government and NGOs staff) to conduct their own appraisal and analysis of open defecation (OD) and take their own action to become open defecation free (ODF).

In Mali, the Open Defecation Free (ODF) status has been defined as follows: "each family has a latrine equipped with a cover that limits the proliferation of flies from the pits; all members of the family exclusively use such latrine to defecate; each latrine is equipped with a hand washing device (water + soap / water + ash bucket)".

To estimate the causal effect of CLTS the researchers need to construct a valid counterfactual in order to calculate what would have happened in the absence of the intervention. Random allocation ensures that on average, treated and untreated communities share the same observables and unobservables. Random assignment to treatment also overcomes the main selection problem found in evaluations, where those who are selected to receive the program may have different attributes than those who were not selected in the first place. These differences can be caused by observable attributes, more wealthy communities, more engaged leaders, better weather, etc, may be more willing to engage in CLTS programs, or by unobservable dimensions too. What is more important is that such differences can be affecting the outcomes the investigators want to measure. Random assignment to the program eliminates selection bias because it ensures that on average, communities receiving the program are similar to the ones that do not receive it.

Although random assignment is at the community level, the basic units of analysis of this evaluation are households. The investigators are interested in health outcomes for children under five, because diarrhea is among the main causes of child mortality. Also, the researchers are interested at looking at morbidity and school attendance for school age children. Finally, improved sanitation is supposed to produce a redistribution in the use of time at the household level. In addition the researchers are very interested at looking at variables that are directly related to the success/failure of the intervention. In particular, the investigators will monitor latrine use, water quality, general hygiene. The team will be able to determine whether lack of impact on health outcomes is due to lack of latrine use despite their availability, or whether it is due to lack of hand hygiene despite use of latrines.

UNICEF has observed in areas where the program has already been implemented that migration is relatively low, so the researchers do not expect much attrition. This decrease in diarrhea can be expected even if the village does not become fully ODF, but take up levels are lower.

The evaluation comprises gathering data at two points in time: a) baseline, before program implementation, b) follow up 12 months after program implementation in order to assess longer-term effects and sustainability. The investigators would be able to gather panel data at the community and at the household level.

While random assignment allows to compare average outcomes across communities, the investigators would also perform multivariate regression analysis in order to improve the precision of our estimates and control for any potential pre-treatment differences. Panel data allows the use of a difference in difference design, if necessary, and also to include initial (before the intervention) characteristics of households and communities. Standard errors will be clustered at the community level.

The communities included in the study understand and agree to be part of the study, meaning that they accept to work on sanitation issues with CLTS either right away or two years later. Randomization will be completed after baseline is conducted. UNICEF and the Directorate of Sanitation of Koulikoro (DNACPN) will conduct the triggering process in the 60 communities assigned to the treatment group.

One of the main concerns of random assignment is the potential contamination of the control group. This happens for example when there are interactions between members of CLTS communities and members of control communities. This is a problem in the presence of shared activities. The problem is that these interactions may cause changes in the control group. At the extreme, control communities and CLTS communities experience the same change, then the researchers will not be able to detect any effect. The researchers will ensure the study communities have geographic buffers, so that interaction is not expected to be very high. In order to check for interaction between family members living in different communities, the team added several questions in the surveys and document the extent of interactions. Another concern that often arises with randomized experiments is that control units may be receiving similar benefits from other interventions. The investigators will monitor control villages to ensure this does not happen and document this aspect of the design.

UNICEF plan to conduct strict monitoring during the intervention period (first 3 months). The research team plans to supplement this work by measuring relevant indicators of intervention compliance during the intervention period and after the end of the intervention.

The investigators will give careful attention to the variation in impacts across different groups, so treatment may be interacted with gender and age indicators, pre-existing characteristics of communities in terms of collective decision-making, among others in order to identify how these factors may explain why some people or some communities gain more than others from the program. Looking at heterogeneity in program impacts also helps in shedding light on the mechanism behind program's success (or failure).

This is one of the first evaluations using impact evaluation techniques with quantitative data [and random assignment] of CLTS programs in the developing world. It will also complement already existing evidence. Another advantage of this evaluation is that it will look carefully at behavioral outcomes that are behind the adoption of better sanitation practices and that are often overlooked in evaluations related to sanitation, which tend to focus more on health outcomes. It is widely accepted that better sanitation improves health, yet there is still much debate over what a cost-effective way to deliver a sanitation intervention may be. Success in delivery will very much depend on whether the program is able to identify bottlenecks that impede adoption of better sanitation practices and whether it is able to solve the issues that are identified.

ELIGIBILITY:
Inclusion Criteria:

* Villages located in rural Mali.
* CLTS targets small villages (less than 4500 inhabitants).
* Open defecation is present

Exclution criteria:

-Villages where CLTS is already in place

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39246 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Diarrhea prevalence of children under five years old | Measured 24 months after the baseline survey (12 months after intervention complete)
  Defined as 3 or more loose or watery defecation events in a 24 hour period. Measured using a 2-day and 2-week recall period.

SECONDARY OUTCOMES:
Length-for-Age Z-scores of children under five years old and children under two years old | Measured 24 months after baseline
  Child's length, standardized to Z-scores using the WHO 2006 growth standards, measured 24 months after baseline.
Stunting Prevalence of children under five years old and children under two years old | Measured 24 months after baseline
  Child's length, standardized to Z-scores using the WHO 2006 growth standards, measured 24 months after baseline. Children with length-for-age Z-scores < - 2 will be classified as stunted.
Weight-for-Age Z-scores of children under five years old and children under two years old | Measured 24 months after baseline
  Child's weight, standardized to Z-scores using the WHO 2006 growth standards, measured 24 months after baseline.
Underweight Prevalence of children under five years old and children under two years old | Measured 24 months after baseline
  Child's weight, standardized to Z-scores using the WHO 2006 growth standards, measured 24 months after baseline. Children with weight-for-age Z-scores < - 2 will be classified as underweight.

OTHER OUTCOMES:
Psychological outcomes: knowledge, risk perceptions, safety, privacy | Measured 24 months after baseline
Community outcomes: level of cooperation and trust, social cohesion, wealth disparities, leadership | Measured 24 months after baseline
  Experimental games can be used to estimate the level of cooperation within communities. A first goal would be to test if and how communication and public exposure of contributions for a public good to the group scrutiny affects the level of cooperation. A public good experiment involves providing endowments to players and asking them to choose how much of their resources to invest in a group project. When making their decision, they know that the experimenter will collect all contributions, double the amount and redistribute it among participants. They are asked to all put their chosen amount in an envelope at the same time and without discussing it. In this situation, no one, except the experimenter, knows how much each of them contributes, but they do know the total contribution. An interesting variation on this game is to let the group members talk before they fill their envelop. Another variation consists in changing the nature of contributions from private to public.
Symptoms of respiratory illness among children under five years old | Measured 24 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maria L. Alzua, Ph.D Econ, Principal Investigator — Universidad Nacional de La Plata
Locations (1):
- Rural Communities in Mali, Bamako, Koulikoro, Mali

REFERENCES:
- [Background] Bernheim Douglas and Antonio Rangel. 2007. Behavioural public economics: welfare and policy analysis with non-standard decision-makers. In Behavioural Economics and its applications. Edited by Peter Diamond and Hannu Vartiainen. Princeton University Press.
- [Background] Bloom, H.S. (1995). Minimum Detectable Effects: A Simple Way to Report the Statistical Power of Experimental Designs. Evaluation Review, 19(5), 547-556.
- [Background] Cardenas, Juan-Camilo. 2003. Real wealth and experimental cooperation: experiments in the field lab. Journal of Development Economics, 70: 263-289.
- [Background] Clasen TF, Bostoen K, Schmidt WP, Boisson S, Fung IC, Jenkins MW, Scott B, Sugden S, Cairncross S. Interventions to improve disposal of human excreta for preventing diarrhoea. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD007180. doi: 10.1002/14651858.CD007180.pub2. PMID 20556776
- [Derived] Pickering AJ, Djebbari H, Lopez C, Coulibaly M, Alzua ML. Effect of a community-led sanitation intervention on child diarrhoea and child growth in rural Mali: a cluster-randomised controlled trial. Lancet Glob Health. 2015 Nov;3(11):e701-11. doi: 10.1016/S2214-109X(15)00144-8. PMID 26475017